CLINICAL TRIAL: NCT07139756
Title: Deciphering the Mechanisms of Central Blood Pressure Regulation in Patients With Parkinson Disease Associated With Orthostatic Hypotension: A 2-phase Observational Study With Healthy Participants and Patients With Parkinson's Disease
Brief Title: Deciphering the Mechanisms of Central BP Regulation in Patients With PD Associated With Orthostatic Hypotension
Acronym: HYPOPARK
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Ecole Polytechnique Fédérale de Lausanne (Other); University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Gregoire Wuerzner; MD, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Other Study IDs: 2024-01828
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease; Orthostatic Hypotension
Keywords: lower body negative pressure; parkinson disease; orthostatic hypotension
MeSH Terms: conditions — Parkinson Disease; Hypotension, Orthostatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Simple blood count, creatinine, sodium, potassium, fasting glucose, pregnancy test for women with childbearing potential
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy volunteers: Healthy volunteers with normal office blood pressure (<140/90 mmHg).
  Lower body negative pressure during brain BOLD fMRI in 3T and 7T MRI scanner.
  Interventions: Diagnostic Test: Lower body negative pressure
- Parkinson patients without orthostatic hypotension: Patients with clinically established Parkinson disease, treated by dopamine replacement therapy, and without orthostatic hypotension as shown by a Schellong test.
  Lower body negative pressure during brain BOLD fMRI, renal contrast-enhanced ultrasound
  Interventions: Diagnostic Test: Lower body negative pressure
- Parkinson patients with orthostatic hypotension: Patients with clinically established Parkinson disease, treated by dopamine replacement therapy, and having orthostatic hypotension as shown by a Schellong test.
  Lower body negative pressure during brain BOLD fMRI, renal contrast-enhanced ultrasound
  Interventions: Diagnostic Test: Lower body negative pressure

INTERVENTIONS:
Diagnostic Test: Lower body negative pressure — LBNP is a technique that redistributes blood from the upper body to the dependent regions of the legs, thus reducing central venous pressure and venous return and thereby activating the sympathetic nervous system (SNS). The subject is placed in a cylindrical airtight tank, which is sealed at the level of the iliac crests, and sub-atmospheric pressure is produced using a vacuum pump. It can be used to characterize the cardiovascular responses to orthostatic stress

SUMMARY:
Phase 1 objective: test the feasibility of using a 3Tesla MRI scanner instead of a 7Tesla MRI scanner to measure brainstem responses to LBNP in healthy participants.

Phase 2 primary objective: compare the brainstem responses to LBNP in patients with PD associated with OH to PD patients without OH using BOLD fMRI

DETAILED DESCRIPTION:
Phase 1 objective: test the feasibility of using a 3Tesla MRI scanner instead of a 7Tesla MRI scanner to measure brainstem responses to LBNP in healthy participants using BOLD fMRI

Phase 2 primary objective: compare the brainstem responses to LBNP in patients with PD associated with OH to PD patients without OH using BOLD fMRI

Phase 2 secondary objectives:

* assess modulation of functional connectivity in response to LBNP (effective connectivity analysis by psycho-physiological interactions (PPI)) and determine differences between the two groups
* assess functional connectivity in resting state and determine differences between the two groups
* compare structural connectivity in both groups using tractography
* compare renal response to LBNP in both groups using contrast-enhanced ultrasound
* compare pre-cerebral flow response to LBNP in both groups

ELIGIBILITY:
Phase 1:

Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 years and <75 years
* Normal office blood pressure (<140/90 mmHg)
* For women of childbearing potential: using or willing to use during the study a reliable contraception method compatible with MRI

Exclusion Criteria:

* Schellong test showing OH (drop of Systolic BP >20 mmHg or Diastolic BP >10 mmHg)
* Pregnant or lactating women
* Refusal to be informed of incidental findings
* Any medication (acute or chronic prescription) except oral contraception
* Clinical significant abnormal blood test as assessed by the investigator
* Chronic or acute illness
* Concomitant participation in a clinical trial
* Blood donation in the 60 previous days
* Contra-indications for MRI
* Unable to follow study procedures
* Having a hierarchical relationship with the investigator or being family of the investigator

Phase 2:

Inclusion Criteria:

* Signed informed consent
* Fulfilling Movement Disorder Society clinical criteria for "clinically established PD"
* Age ≥18 years and <75 years
* PD treated by dopamine replacement therapy (DRT)
* Willing and able to comply with the visit schedule and study procedures
* Autonomous in daily life
* Schellong test showing OH (drop of Systolic BP >20 mmHg or Diastolic BP >10 mmHg)(for study group with OH) or no OH (for studygroup without OH)
* For women of childbearing potential: using or willing to use during the study a reliable contraception method compatible with MRI

Exclusion Criteria:

* Unable to give an informed consent
* BP > 180/110 mmHg on 24-hour ambulatory blood pressure monitoring
* eGFR < 45 ml/min/1.73 ml/min/m2 by CKD-EPI equation
* having contra-indications for MRI
* Pregnant or lactating women
* Refusal to be informed of incidental findings
* Allergy to components of contrast agent Sonovue®
* Living in an institution
* Dementia
* Type 2 diabetes
* Stroke or myocardial infarction in the past 6 months
* Blood donation in the previous 6 months
* Active oncology treatment
* Having a hierarchical relationship with the investigator or being family of the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Phase 1: population of healthy participants Phase 2: population of PD patients with or without OH
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Differences and changes in BOLD fMRI signal intensity | 1.5 hour
  Changes in brain BOLD fMRI signal in the dorsolateral medulla of the brainstem in response to LBNP

SECONDARY OUTCOMES:
Functional connectivity | 1.5 hour
  Activation patterns in spatially separated brain regions tending to have synchronous activity in resting state and activation pattern change during LBNP
Structural connectivity | 30 minutes
  Map of anatomical (neural) connections within the brain in PD patients with and without OH
Contrast-enhanced renal ultrasound | 1.5 hour
  Changes in renal perfusion in response to LBNP
pre-cerebral blood flow | 30 minutes
  changes in pre-cerebral blood flow in response to LBNP

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire Wuerzner, Principal Investigator — CHUV
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: one year after publication of the data